CLINICAL TRIAL: NCT00690729
Title: Cognitive-Behavioral Treatment of Obsessive Compulsive Disorder in Children and Adolescents
Brief Title: Cognitive-Behavioral Bibliotherapy for the Treatment of Obsessive Compulsive Disorder in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Kimberli Treadwell/Assistant Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H06-170
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2010-08

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Bibliotherapy - cognitive behavior therapy focusing on exposure and response prevention directed by the family
  Interventions: Behavioral: Cognitive Behavioral Bibliotherapy
- 2 (Active Comparator): Cognitive Behavioral Therapy - therapist-directed exposure response prevention over a 12-week period
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Bibliotherapy — Minimal therapist direction for self-guided bibliotherapy involving exposure and response prevention
  Arms: 1
Behavioral: Cognitive Behavioral Therapy — Therapist-directed exposure and response prevention
  Arms: 2

SUMMARY:
This 16-week program examines cognitive behavioral bibliotherapy to typical therapist-directed cognitive behavior therapy for children and adolescents with Obsessive Compulsive Disorder.

DETAILED DESCRIPTION:
This study is designed to compare self-directed bibliotherapy and therapist-directed cognitive behavioral therapy for children and adolescents with Obsessive Compulsive Disorder (OCD). Both treatments involve exposure and response prevention (EX/RP), in which the child confronts OCD fears and is asked to refrain from compulsive rituals (such as repetitive handwashing, counting, etc.). Participants are requested to complete an initial evaluation to determine diagnosis, and four follow-up evaluations to assess symptom severity and change due to treatment for a total of 16 weeks. Participant involvement to self-directed bibliotherapy versus traditional cognitive-behavioral treatment will be determined through random assignment.

In the bibliotherapy condition, the child or adolescent will meet with a therapist twice over the course of treatment, along with a parent. The therapist will discuss a self-directed program of EX/RP to be implemented at a pace deemed appropriate by child and parent at their own home. The child and parent will be provided with a manual designed to instruct them how to cope with Obsessive Compulsive Disorder. This treatment involves the parent and child reading the book, performing exercises, and monitoring symptoms on a weekly basis for 8 weeks.

In the therapist-directed treatment condition, the child or adolescent will meet weekly with a therapist along with their parent. The therapist, parent, and child will work together to design and implement a program of EX/RP. This treatment involves performing exercises, monitoring symptoms on a weekly basis, and completing homework assignments. Parents will be asked to help coach their child with at-home exercises challenging the Obsessive Compulsive Disorder. This treatment lasts 12 weeks.

Evaluations will be conducted following the completion of each treatment to assess the efficacy of each treatment on OCD symptoms. The treatment and evaluations for OCD are provided free of charge.

ELIGIBILITY:
Inclusion Criteria:

* Ages 8-18 years old
* Primary diagnosis of Obsessive Compulsive Disorder
* Both parent and child fluent in English
* Parents must read at least a 7th grade reading level

Exclusion Criteria:

* Primary psychiatric diagnosis other than OCD
* Current threat of harm to self or others
* New use or dosage change of OCD medication 60 days prior to starting program
* Current involvement with another psychosocial therapy

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2005-07; Primary Completion 2010-03 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Child Yale-Brown Obsessive Compulsive Scale | 12 weeks

SECONDARY OUTCOMES:
NIMH Clinician's Global Impression | weeks 4, 8, 12, 16
Children's Obsessional Compulsive Inventory | weeks 4, 8, 12, and 16
Child OCD Impact Scale | weeks 4, 8, 12, 16
March Anxiety Scale for Children | weeks 4, 8, 12, 16
Children's Depression Inventory | weeks 4, 8, 12, 16
Child Behavior Checklist | weeks 4, 8, 12, 16
Family Assessment Measure III | weeks 4, 8, 12, 16

CONTACTS AND LOCATIONS:
Overall Officials: Kimberli Treadwell, Ph.D., Principal Investigator — University of Connecticut
Locations (4):
- United States (4):
  - Institute of Living, Hartford, Connecticut
  - University of Connecticut, Storrs, Connecticut
  - University of Connecticut, Waterbury, Connecticut
  - University of Connecticut, West Hartford, Connecticut